CLINICAL TRIAL: NCT05690828
Title: Etude e-ONCOGITE : Évaluation d'Une Prise en Charge Cognitive adaptée au " Chemobrain" Chez Des Patientes traitées Pour un Cancer de Sein.
Brief Title: Evaluation of Cognitive Management for Chemobrain in Patients Treated for Breast Cancer.
Acronym: e-ONCOGITE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Bergonié (Other)
Collaborators: University of Bordeaux (Other); Association Oncogite (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IB2022-04
Record Dates: First submitted 2023-01-10; First posted 2023-01-19 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Breast Cancer
Keywords: Cognition
MeSH Terms: conditions — Breast Neoplasms | interventions — Cognitive Remediation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Cognitive remediation) (Experimental)
  Interventions: Behavioral: Cognitive remediation
- Group 2 (No cognitive remediation) (No Intervention)

INTERVENTIONS:
Behavioral: Cognitive remediation — The cognitive remediation programme shall be run either in video workshops or face to face workshops and in home sessions via a web app. The programme will run for 4 months during which there will be 3 different evaluations. A first evaluation after randomisation, a second evaluation 4 months after inclusion (corresponding to the end of the programme), and a third evaluation 8 months after inclusion for the experimental group (4 months after the end of the programme). The face to face workshops will take 8 to 10 participants and will be led by a neuropsychologist.
  Arms: Group 1 (Cognitive remediation)

SUMMARY:
This project will investigate the efficacy of a cognitive remediation programme in patients treated for breast cancer. patients will be randomized between "no intervention" and "intervention programme". Efficay will be assessed in term of improved quality of life.

DETAILED DESCRIPTION:
Medical progress in the treatment of cancer has prolonged patients' life expectancy. This improvement has led researchers to become concerned about the long-term negative effects of cancer treatments on quality-of-life. In particular, previous studies have identified complaints that have been submitted concerning the cognitive status of patients treated with chemotherapy (Berglund et coll., 1991). All of these cognitive changes are collectively grouped under the term chemobrain.

The consequences of treatments remain however underestimated, as the priority when diagnosing cancer remains the patient's short- to medium-term survival; yet, quality-of-life contributes to the long-term survival of patients (Kramer, 2000).

In addition to medical treatments, psychosocial care adapted to the specific needs of subjects is thus important for improving their quality-of-life and helping them return to work. Even if initiatives have multiplied over the past few decades in the psychosocial management of these subjects (e.g., supportive care), that related to cognitive disorders in subjects having survived cancer remains a little documented field. Cognitive deficiency in cancer survivors is said to be moderate (Razaq et coll., 2017), which makes survivors ideal candidates for cognitive rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged 20 to 60 years inclusive.
2. Localised breast cancer having required neoadjuvant or adjuvant chemotherapy, the last cycle of which took place between 2 and 24 months prior to inclusion.
3. Informed consent dated and signed.
4. Patient with French social security cover in accordance with French law on biomedical research (Article 1121-11 of the French code of public health).

Exclusion Criteria:

1. Metastatic breast cancer.
2. Presence of unstable psychiatric or neurological disorders likely to affect cognition (information requested directly from the participant)
3. History of drug abuse.
4. Patient who cannot read or understand French.
5. Patient already included in this study.
6. Patient having participated in onCOGITE workshops.
7. Patient participating in another clinical trial evaluating cognitive remediation.
8. Patient deprived of freedom or subject to legal protection measures (under guardianship, in custody of the court, or family-member guardianship order).

Ages: 20 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 164 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with improved quality of life (Emotional and functional QoL) | 4 months after initiation of the cognitive stimulation protocol using the "onCOGITE" method
  Improved QoL is defined as a significant improvement (i.e. at least a 3-point increase of the total score) in both the Emotional Well-Being (EWB) and Functional Well-Being (FWB) subscales of the FACT-B self-questionnaire (Functional Assessment of Cancer Therapy -Breast - Brady et al. J Clin Oncol 1997).

SECONDARY OUTCOMES:
Number of participants with improved quality of life (physical QoL) | 4 months after initiation of the cognitive stimulation protocol using the "onCOGITE" method
  Improved QoL is defined as a significant improvement (i.e. at least a 3-point increase of the total score) in the physical Well-Being subscale of the FACT-B self-questionnaire (Functional Assessment of Cancer Therapy -Breast - Brady et al. J Clin Oncol 1997).
Number of participants with improved quality of life (Social/family QoL) | 4 months after initiation of the cognitive stimulation protocol using the "onCOGITE" method
  Improved QoL is defined as a significant improvement (i.e. at least a 3-point increase of the total score) in the Social/family subscale of the FACT-B self-questionnaire (Functional Assessment of Cancer Therapy -Breast - Brady et al. J Clin Oncol 1997).

CONTACTS AND LOCATIONS:
Overall Officials: Véronique GERAT-MULLER, PhD, Principal Investigator — v.gerat-muller@bordeaux.unicancer.fr
Locations (1):
- Institut Bergonié, Comprehensive Cancer Center, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No